CLINICAL TRIAL: NCT01531920
Title: A Phase 1 Study in Healthy Subjects to Determine the Safety, Tolerability, Psychomotor Function and Cognitive Effects of Perampanel When Administered With Alcohol
Brief Title: A Study in Healthy Subjects to Determine the Effects When Alcohol is Administered With Perampanel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2007-E044-030
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-01

CONDITIONS: Central Nervous System
MeSH Terms: interventions — Ethanol; perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- alcohol + placebo (Other): Part A alcohol + placebo
  Interventions: Drug: alcohol + placebo
- alcohol + perampanel (Other): Part A : alcohol + perampanel
  Interventions: Drug: alcohol + perampanel
- perampanel + alcohol (Other): Part B: perampanel + alcohol
  Interventions: Drug: perampanel + alcohol
- placebo + alcohol (Other): Part B: placebo + alcohol
  Interventions: Drug: placebo + alcohol

INTERVENTIONS:
Drug: alcohol + placebo — Part A alcohol + placebo
  Arms: alcohol + placebo
Drug: alcohol + perampanel — Part A: alcohol + perampanel
  Arms: alcohol + perampanel
Drug: perampanel + alcohol — Part B: perampanel + alcohol
  Arms: perampanel + alcohol
Drug: placebo + alcohol — Part B: placebo + alcohol
  Arms: placebo + alcohol

SUMMARY:
A Phase 1 study in healthy subjects to determine the safety, tolerability, psychomotor function, and cognitive effects of perampanel when administered alone and with alcohol.

ELIGIBILITY:
Inclusion:

* Healthy male and female subjects
* Females agreed to use two medically acceptable methods of contraception, unless they were surgically sterile
* Aged 18-55 yrs, inclusive
* Achieved a Continuous Tracking Test (CTT )score increase of >1.5 pixels from pre-alcohol when dosed with alcohol during the Screening Period (Day minus 8 plus/minus 2 days)
* Had a current driving license and drove regularly (e.g., more than 1000 miles a year (Part B only)

Exclusion:

* Any history of significant alcohol abuse or psychiatric disease, requiring inpatient admission or prolonged treatment with psychotropic medication
* Unable to follow the instructions for the psychometric testing
* Intolerant to the driving simulator (Part B only)
* Unable to adhere to long periods of confinement (subjects who could not follow the instructions of the protocol, including the meals)
* Use of prescription drugs or over-the-counter (OTC) medications within 2 weeks prior to Screening (unless drug had a long half life [i.e., 5 x t 1/2>2 weeks]) with the exception of paracetamol (up to 4 g/day), which was allowed up to 12 hours prior to dosing
* Had taken any inhibitor of CYP450 within 2 weeks prior to the first dosing (e.g., grapefruit, grapefruit juice, grapefruit-containing beverages, or Seville orange products)
* Had taken St John's Wort or other dietary aids known to induce CYP3A4 within 4 weeks prior to dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Part A: Changes on Psychomotor Performance (Continuous Tracking Test [CTT]), due to perampanel and alcohol combined and perampanel alone | baseline to Part A Day 1
Part B: Changes on Psychomotor Performance (Continuous Tracking Test [CTT]) due to perampanel and alcohol combined and perampanel alone | baseline to Part B Day 62
Part B:Changes in Cognitive Function due to perampanel and alcohol combined and perampanel alone | baseline to Part B Day 62
Part B: Part B: Changes in driving performance (simulated) due to perampanel and alcohol combined and perampanel alone | Part B Day 34

SECONDARY OUTCOMES:
Part A: Incidence of AEs when perampanel is administered in combination with alcohol | baseline to Part A Day 29
Part B: Incidence of AEs when perampanel is administered in combination with alcohol | baseline to Part B Day 62

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Bendel, Principal Investigator — Surrey Clinical Research Centre
Locations (1):
- Guildford, United Kingdom